CLINICAL TRIAL: NCT04566965
Title: Serology to Covid for Recording Exposures and Evaluating Needs (SCREEN)
Brief Title: Serology to COVID-19 for Recording Exposures and Evaluating Needs
Acronym: SCREEN
Status: Terminated | Type: Observational
Why Stopped: CARES and institutional funding ended
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: SCREEN
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Coronavirus; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serial collections of weekly self-collected nasal swabs and monthly blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full-Time CCHMC Employees: All CCHMC full-time residents and fellows who have some direct contact with patients and their families as part of normal workplace duties.
  Interventions: Diagnostic Test: SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 — 1. Testing weekly samples from nasal swabs to promptly diagnose acute COVID-19 infection.
  2. Testing monthly serum samples to document post-viral infection.

SUMMARY:
As the global and pandemic spread of the novel coronavirus (SARS-CoV-2, COVID-19) continues, many knowledge gaps remain with regard to the epidemiology and transmission of infection, as well as the normal immunological responses after viral exposure. Cincinnati had its first confirmed case of COVID-19 on March 14, 2020, and despite extensive shelter-in-place and social distancing efforts, community spread continues at over 150-200 new cases per week. As new residents and fellows arrive in July 2020 to Cincinnati Children's Hospital Medical Center (CCHMC), many of whom come from metropolitan areas across the country, it is imperative that investigators determine the current prevalence of infection, measure the cumulative incidence of infection over the next 12-24 months, investigate the normal antibody patterns after infection, and help elucidate what constitutes a protective immunological response. The investigators have a unique but time-limited opportunity to optimally track the epidemiology and natural history of SARS-CoV-2 infection among trainees at CCHMC, including risk factors for transmission and immunological recovery. SCREEN will investigate epidemiological and immunological features of SARS-CoV-2 virus infection within the cohort of CCHMC residents and fellows who have patient contact. By collecting and analyzing weekly serial samples for SARS-CoV-2 (nasal swab for virus by PCR) and monthly serological exposure (serum antibodies by ELISA), the investigators will determine the prevalence and cumulative incidence of infection by SARS-CoV-2; the investigators will also document the antibody responses over time and identify cases of apparent viral recrudescence or re-infection.

ELIGIBILITY:
Inclusion Criteria:

* Current full-time residents and fellows at CCHMC
* Cell phone that can be used for text messaging or web-based viewing of surveys
* Willing and able to provide informed consent
* Ability to comply with all study related evaluations and follow-up

Exclusion Criteria:

* Any condition or illness that makes study participation ill-advised

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult men and women who are CCHMC full-time residents and fellows who have some direct contact with patients and their families as part of normal workplace duties.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The 12-month cumulative incidence of acquired COVID infection in the study cohort. | Weekly for 12 months
  Acquired COVID is defined as testing negative for COVID at baseline and having 1 or more weekly nasal swab samples testing positive for the virus by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Mary Allen Staat, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sue Poynter Wong, MD, MEd, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No